CLINICAL TRIAL: NCT07132580
Title: The Effect of Bright Light Therapy on Sleep Quality, Cancer-Related Fatigue, and Emotional Symptoms in Gynecologic Cancer Survivors: A Randomized Controlled Trial
Brief Title: Effects of Bright Light on Sleep Quality, Fatigue , and Mood Symptoms in Survivors With Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202400345A3C601; IRB Protocol ID (Other: 202400345A3C601)
Record Dates: First submitted 2025-08-10; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Gynecologic Cancer Survivors; Sleep Quality; Fatigue; Mood Symptoms
Keywords: light therapy; gynecologic cancer; chemotherapy; sleep quality; fatigue; emotional symptoms
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the bright light group or the dim red light control group in a parallel design. Each participant received only one type of light intervention throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright Light Intervention Group (Experimental): Participants in this group received daily morning exposure to bright white light (506 lux) using the Re-Timer® light therapy glasses for 45 minutes per day, over a 4-week period.
  Interventions: Device: Re-Timer® light therapy glasses
- Usual Care (Other): Participants in this group received usual care and did not receive any light therapy intervention during the study period.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Re-Timer® light therapy glasses — Participants wore Re-Timer® glasses that emitted bright white light at 506 lux for 30 minutes each morning, over a 4-week intervention period.
  Arms: Bright Light Intervention Group
Other: Usual Care — Participants received standard follow-up care with no light therapy intervention during the 4-week period.
  Arms: Usual Care

SUMMARY:
Objective: This study aimed to examine the efficacy of light therapy in improving sleep quality, reducing fatigue, and alleviating emotional symptoms among patients diagnosed with gynecologic cancer.

Methods: A randomized controlled trial was conducted at a medical center in northern Taiwan. Inclusion criteria included patients aged 18 years or older with a physician-confirmed diagnosis of gynecologic cancer and a score of ≥ 9 on the Chinese version of the Insomnia Severity Index (ISI-C). Eligible participants were randomly assigned to an experimental group or a control group (each with 47 subjects). At baseline (T0), all participants completed a demographic and treatment questionnaire, the ISI-C, the Taiwan version of the Brief Fatigue Inventory (BFI-T), and the Distress Thermometer (DT). The experimental group then underwent daily light therapy sessions via a circadian regulator for 30-40 minutes within 30 minutes of waking for four weeks. Meanwhile, the control group continued their usual routines during the same period. Follow-up assessments were conducted on days 7 (T1), 14 (T2), 21 (T3), and 28 (T4) post-intervention. Data was analyzed using SPSS 26.0, and generalized estimating equations (GEE) were employed to assess the effectiveness of light therapy.

Results: Generalized Estimating Equations (GEE) will be applied to examine group differences over time in sleep quality, fatigue, and emotional symptoms, in order to assess the effects of the intervention.

Conclusion: Light therapy is proposed as a potentially safe, low-risk, and cost-effective non-pharmacological intervention for improving sleep quality, reducing fatigue, and alleviating emotional distress in patients with gynecologic cancer following chemotherapy. This study is designed to evaluate the feasibility and potential effects of light therapy in this population, with the goal of informing future clinical applications.

DETAILED DESCRIPTION:
Background and Rationale

Survivors of gynecologic cancers often experience persistent sleep disturbances, cancer-related fatigue, and emotional distress even after treatment has ended. These symptoms can significantly affect daily functioning, emotional well-being, and overall quality of life. Bright light therapy (BLT), a non-pharmacological intervention, has been shown in other populations to help regulate circadian rhythms and improve sleep and fatigue by suppressing melatonin levels. However, the application of BLT in gynecologic cancer survivors has not been well studied. This trial is designed to explore the potential of BLT in addressing these symptoms in this specific population.

Objectives

The primary objective is to evaluate the effects of a four-week bright light therapy intervention on sleep quality, fatigue, and emotional symptoms among gynecologic cancer survivors. It is hypothesized that participants receiving BLT will demonstrate improved outcomes in these domains compared to those receiving usual care.

Study Design

This is a randomized, controlled, single-blind trial with a parallel-group design. Eligible participants will be randomly assigned in a 1:1 ratio to either the intervention group (BLT) or the control group. Outcome assessors will remain blinded to group allocation throughout the study.

Intervention

Participants in the intervention group will receive bright light therapy using Re-Timer® light therapy glasses, which emit green-blue light at an intensity of 506 lux. Participants will be instructed to wear the glasses for 45 minutes each morning over four consecutive weeks. Sessions are self-administered at home between 7:00 AM and 9:00 AM, based on circadian rhythm guidance.

Control Condition

The control group will receive usual care and will not be provided with any light therapy. Participants in this group will be instructed to maintain their typical daily routines and avoid introducing new interventions that could impact sleep or mood during the study period.

Outcome Measures and Timepoints

Outcome data will be collected through an online questionnaire via the LINE messaging app at the following timepoints:

T1: Day 7 of intervention

T2: Day 14 of intervention

T3: Day 21 of intervention

T4: Day 28 of intervention

The following instruments will be used:

Insomnia Severity Index - Chinese version (ISI-C): to assess insomnia symptoms

Brief Fatigue Inventory - Taiwanese version (BFI-T): to assess cancer-related fatigue

Distress Thermometer (DT): to assess emotional distress

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged 18 years or older.
2. Diagnosed with ovarian cancer, cervical cancer, fallopian tube cancer, or endometrial cancer, and have completed primary treatment (surgery, chemotherapy, or radiation) for more than 3 months, Currently in the treatment stage.
3. Insomnia Severity Index-Chinese Version (ISI-C) score ≥ 9, indicating clinical insomnia (Yang et al., 2009).
4. If currently using psychiatric medications, the dosage must have remained stable for at least 6 weeks prior to participation.
5. Able to speak Mandarin or Taiwanese fluently and read and write in Chinese.
6. Able to use a smartphone.
7. Conscious, capable of understanding the study procedures, willing to sign informed consent, and agree to participate.

Exclusion Criteria:

1. History of psychiatric hospitalization or severe psychiatric disorders within the past 6 months.
2. Eye diseases or ophthalmologic surgery within the past two weeks, conditions contraindicating light therapy, or use of photosensitizing drugs (e.g., cataracts).
3. Currently taking hypnotic medications.
4. Habitual smoking or alcohol use.
5. Working night shifts, rotating shifts, or frequent travel across multiple time zones.
6. Currently pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index - Chinese version (ISI-C) | Day 7 (T1), Day 14 (T2), Day 21 (T3), and Day 28 (T4) after intervention start.
  To evaluate the change in insomnia severity before and after the intervention using the Insomnia Severity Index - Chinese version (ISI-C). Higher scores indicate more severe insomnia.

SECONDARY OUTCOMES:
Cancer-related fatigue (BFI-T) | Day 7 (T1), Day 14 (T2), Day 21 (T3), and Day 28 (T4) after the start of the intervention.
  To assess the level of cancer-related fatigue using the Brief Fatigue Inventory - Traditional Chinese version (BFI-T).
  The BFI-T includes 9 items rated on a 0-10 numeric scale, with higher scores indicating greater fatigue severity and interference.
Emotional distress (Distress Thermometer, DT) | Day 7 (T1), Day 14 (T2), Day 21 (T3), and Day 28 (T4) after the start of the intervention.
  To measure overall emotional distress using the Distress Thermometer (DT), a single-item visual analog scale ranging from 0 (no distress) to 10 (extreme distress).
  Participants indicate their distress levels during the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Lingya Hsu, MSN, RN, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this article will be shared. The shared data will include the variables analyzed for primary and secondary outcomes, baseline characteristics, and adverse events (if applicable).
  Data will be available upon reasonable request to qualified researchers for the purpose of academic and non-commercial use. Interested researchers must provide a methodologically sound proposal and obtain approval from the principal investigator and the Institutional Review Board (IRB) of the host institution.
  Data will be available starting 6 months after publication of the study results and will remain available for up to 3 years.
  Requests for data sharing should be submitted to the corresponding author via email.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be available beginning 6 months after publication of the study results. Data will remain available for 3 years and may be extended upon request and approval by the principal investigator.
Access Criteria: Qualified researchers affiliated with academic or non-profit institutions may request access to individual participant data (IPD) and supporting documents (e.g., protocol, informed consent form, analytic code) for the purpose of scientific research. Requests must include a detailed research proposal and be submitted to the principal investigator for review and approval. Data will be de-identified to protect participant confidentiality, and access will be granted through a secure data sharing platform.

REFERENCES:
- [Background] Lin LY, Tam KW, Huang TW. Effect of bright light therapy on cancer-related fatigue and related symptoms: A systematic review and meta-analysis of randomized controlled trials. J Psychosom Res. 2023 Nov;174:111501. doi: 10.1016/j.jpsychores.2023.111501. Epub 2023 Sep 27. PMID 37797569
- [Background] Fox RS, Baik SH, McGinty H, Garcia SF, Reid KJ, Bovbjerg K, Fajardo P, Wu LM, Shahabi S, Ong JC, Zee PC, Penedo FJ. Feasibility and Preliminary Efficacy of a Bright Light Intervention in Ovarian and Endometrial Cancer Survivors. Int J Behav Med. 2021 Feb;28(1):83-95. doi: 10.1007/s12529-020-09861-0. PMID 32080797
- [Background] Ozerdogan N, Ozkaraman A, Tuncer Yilmaz B, Oge T, Yalcin OT. The Effect of Bright White Light on Fatigue Levels in Patients with Gynecological Cancer: A Randomized Control Trial. J Palliat Care. 2023 Oct;38(4):416-423. doi: 10.1177/08258597221127795. Epub 2022 Sep 25. PMID 36154518
- See also: Cancer Statistics - Ministry of Health and Welfare Taiwan — https://www.hpa.gov.tw/Pages/List.aspx?nodeid=269
- See also: NCCN Distress Thermometer - Traditional Chinese — https://www.nccn.org/professionals/physician_gls/pdf/distress_tool_chinese_traditional.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT07132580/Prot_SAP_000.pdf